CLINICAL TRIAL: NCT00896727
Title: Prediction of Therapeutic Response Using AQUA™ Quantitative Protein Expression Analysis of ER, PgR, and HER2 of Breast Cancer Tissue Microarrays From SWOG Protocol 9313
Brief Title: S9313A Protein Expression Analysis of Breast Cancer Tissue Microarrays From Clinical Trial SWOG-9313
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000467801; SWOG-S9313-INT-0137-ICSC (Other: SWOG); NCI-2009-00806 (Other: NCI)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gene Expression Profiling; Fluorescent Antibody Technique

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: protein expression analysis
Other: fluorescent antibody technique
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying the proteins expressed in tumor tissue samples in the laboratory from patients with cancer may help doctors learn more about biomarkers related to cancer. It may also help doctors predict how patients respond to treatment.

PURPOSE: This laboratory study is looking at protein expression in predicting response to treatment using tumor tissue samples from women with stage I, stage II, or stage IIIA breast cancer treated on clinical trial SWOG-9313.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess in-situ protein expression of estrogen receptor (ER), progesterone receptor (PR), HER-2, and p53 by automated quantitative analysis (AQUA™) and multiplexed analysis at 2 markers per slide using tumor tissue from women with stage I, stage II, or stage IIIA breast cancer treated on clinical trial SWOG-9313.
* Assess the main effects of ER, PR, HER-2, and p53, as well as interactions to generate classes formed by clustering of biomarkers, on a large breast cancer tissue microarray to predict disease-free and overall survival of patients who received high-dose cyclophosphamide and doxorubicin hydrochloride on clinical trial SWOG-9313.

OUTLINE: This is a multicenter study. Patients are stratified according to receptor status and menopausal status.

Tumor tissue samples are analyzed by quantitative protein expression analysis (AQUA™, a fluorescent antibody technique) for estrogen receptor, progesterone receptor, p53 and HER-2. AQUA™ is used to assess markers individually and as ratios with the use of clustering algorithms to define reproducible classifications of tissue from patients treated on SWOG-9313 as a function of molecular classification.

Results of the AQUA™ testing are compared to immunohistochemistry and fluorescent in situ hybridization (FISH) results obtained on SWOG-9313.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of primary invasive adenocarcinoma of the breast

  * Stage I-IIIA disease (T1-3, N0-1, M0)
* Enrolled on clinical trial SWOG-9313
* Tumor tissue available for testing

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from SWOG 9313 consented to banking
Sampling Method: Non-Probability Sample
Enrollment: 2100 (Actual)
Dates: Start 2006-07-17 (Actual); Primary Completion 2009-01-02 (Actual); Study Completion 2009-04-02 (Actual)

PRIMARY OUTCOMES:
In-situ protein expression of estrogen receptor (ER), progesterone receptor (PR), HER-2, and p53 as measured by automated quantitative analysis (AQUA™) | Retrospectively at baseline
  at baseline
Main effects of ER, PR, HER-2, and p53, as well as interactions to generate classes formed by clustering of biomarkers, on a large breast cancer tissue microarray to predict disease-free and overall survival | Retrospectively at baseline
  at baseline

CONTACTS AND LOCATIONS:
Overall Officials: David Rimm, MD, Principal Investigator — Yale University
Locations (1):
- Yale Cancer Center, New Haven, Connecticut, United States